CLINICAL TRIAL: NCT05900596
Title: Fetal Scalp pH During Labour: is it Worth Repeating
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, TOURNIER Mathilde, Resident, Obstetrics and Gynecology, Principal Investigator, Central Hospital, Nancy, France
Other Study IDs: 2023PI036
Record Dates: First submitted 2023-05-26; First posted 2023-06-12 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Abnormal Fetal Heart Rate
Keywords: fetal scalp blood sampling; fetal blood sampling; cesarean section; non-reassuring fetal heart rate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pH < 3: Patients one or two fetal blood sampling
  Interventions: Diagnostic Test: Fetal blood sampling
- pH > 3: Patients with three or more fetal blood sampling
  Interventions: Diagnostic Test: Fetal blood sampling

INTERVENTIONS:
Diagnostic Test: Fetal blood sampling — Fetal scalp blood sampling and analysis

SUMMARY:
In order to reduce the cesarean sections rate, an adjunctive test is recommended in case of non-reassuring fetal heart rate tracing. In France, the reference adjunctive test is fetal scalp blood sampling. However, there is no study about the repetition of fetal blood sampling. Our hypothesis is that the repetition of fetal blood sampling is useful when fetal heart rate stays non-reassuring and may lead to vaginal delivery without impair neonatal prognostic. Therefore, our objective was to compare the patients with three or more fetal blood sampling with the patients with one or two.

ELIGIBILITY:
Inclusion Criteria:

* One fetal blood sampling during labour or more
* Singleton pregnancy
* Gestational age equal or above 37 weeks
* No contra-indication of fetal blood sampling
* No pregnancy complication

Exclusion Criteria:

* Sampling failure
* Incomplete file

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Regional University Maternity of Nancy
Sampling Method: Non-Probability Sample
Enrollment: 130 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Delivery | baseline
  Vaginal delivery, operative delivery, cesarean section

SECONDARY OUTCOMES:
Apgar score | baseline
  value of Apgar score at five minutes of life
umbilical cord pH | baseline
  value of umbilical cord pH
umbilical cord lactates | baseline
  value of umbilical cord lactates
neonatal care intensive unit transfer | baseline
  rate of neonatal care intensive unit transfer

CONTACTS AND LOCATIONS:
Locations (1):
- Regional University Maternity of Nancy, Nancy, Meurthe-et-Moselle, France

IPD SHARING:
Plan to Share IPD: No